CLINICAL TRIAL: NCT00266318
Title: A Phase 4 Open-Label Pilot Study of the Safety and Tolerability of High Dosage of CIFN Plus RBV Administered Daily for 48 Weeks in HCV Genotype 1 Infected Patients Who Are Nonresponders to Prior Pegylated Interferon Alfa Plus RBV Therapy
Brief Title: Study of High Dosage CIFN Plus RBV for HCV Genotype 1 Infected Patients Who Are Nonresponders to Prior Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Collaborators: InterMune (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 164-04
Record Dates: First submitted 2005-12-14; First posted 2005-12-16 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2008-04

CONDITIONS: Hepatitis C
Keywords: Hepatitis C Nonresponder; Genotype 1; Interferon Alfacon-1; Consensus Interferon; CIFN; Infergen; Ribavirin
MeSH Terms: conditions — Hepatitis C | interventions — interferon alfacon-1; Ribavirin

INTERVENTIONS:
Drug: Interferon Alfacon-1 and Ribavirin

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of combination therapy of daily interferon alfacon-1 (Infergen, CIFN) at high dosage (24 mcg) with ribavirin (based on body weight) for 48 weeks in HCV genotype 1 infected subjects, who are non-responders to previous pegylated interferon alfa plus ribavirin therapy.

This is an open-label, multicenter study. All subjects will receive Infergen 24 mcg administered by injection daily plus ribavirin 800-1400 mg (based on body weight) administered by mouth daily for 48 weeks

* If any 5 of the first 10 subjects can not tolerate the 24 mcg daily dosage of Infergen by week 4, as determined by the principal investigator, then the dosage of Infergen will be changed to 15 mcg administered by injection daily plus ribavirin 800-1400 mg (based on body weight) administered by mouth daily for 48 weeks

ELIGIBILITY:
Inclusion Criteria:

* Must have documented failure to respond to past treatment with a Pegylated IFN + RBV. Failure to respond to past treatment is defined as positive HCV RNA at 12 weeks and less than a 2 log drop from baseline; OR positive HCV RNA and greater than 2 log drop from baseline at week 12 and must have received 24 weeks of therapy and still have a positive HCV RNA
* Must have tolerated previous hepatitis C therapy
* Must be off hepatitis C therapy for 3 months prior to study participation
* Must have had a liver biopsy within the past 5 years

Exclusion Criteria:

* Decompensated liver disease
* Laboratory abnormalities as per protocol
* HIV+
* Autoimmune disease
* Unstable or deteriorating cardiovascular or cerebrovascular disease
* History of seizures in past 5 years
* Alcohol or drug abuse in past year
* Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-12; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
*Assessment of safety and tolerability of high dosage Infergen plus ribavirin including adverse events;study medication dose reduction, interruptions, and discontinuations; and BDI-II scores

SECONDARY OUTCOMES:
*Sustained viral response defined as the absence of detectable HCV RNA at week 72

CONTACTS AND LOCATIONS:
Overall Officials: Henry C. Bodenheimer, M.D., Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States

REFERENCES:
- [Background] Cornberg M, Hadem J, Schuppert F, Reiser M, Schmidt H, Marschal O, et al. 2002. Retreatment of hepatitis C nonresponder patients with consensus interferon and ribavirin: a randomized controlled multicenter study. Hepatology 36(4 pt 2): 575A.
- [Result] Barbaro G, Barbarini G. Consensus interferon for chronic hepatitis C patients with genotype 1 who failed to respond to, or relapsed after, interferon alpha-2b and ribavirin in combination: an Italian pilot study. Eur J Gastroenterol Hepatol. 2002 May;14(5):477-83. doi: 10.1097/00042737-200205000-00003. PMID 11984144
- [Result] da Silva LC, Bassit L, Ono-Nita SK, Pinho JR, Nishiya A, Madruga CL, Carrilho FJ. High rate of sustained response to consensus interferon plus ribavirin in chronic hepatitis C patients resistant to alpha-interferon and ribavirin: a pilot study. J Gastroenterol. 2002;37(9):732-6. doi: 10.1007/s005350200119. PMID 12375147
- [Result] Buggisch P, Seegers B, Hinrichsen H, Hueppe D, Reiser M, de Heer G, et al. 2002. Combination treatment with consensus-interferon and ribavirin for chronic hepatitis C patients with non-response relapse to previous treatment with alpha-interferon and ribavirin. Hepatology 36 (4 pt 2): 363A.
- [Result] Hass HG, Nehls O, Gregor M, Kaiser S, Kreysel C. Treatment of chronic hepatitis C in naive patients with high-dose interferon-alpha2a induction therapy and two different ribavirin doses. Dig Liver Dis. 2004 May;36(5):367-8. doi: 10.1016/j.dld.2004.01.009. No abstract available. PMID 15191208
- [Result] Kaiser S, Hass H, gregor M. 2002B. High viral response rates in previous interferon/ribavirin nonresponder patients with chronic hepatitis C retreated with consensus interferon. Hepatology 36(4 pt 2): 358A.
- [Result] Kaiser S, Hass H, Gregor M. 2003. Successful retreatment of Peginterferon nonresponder patients with chronic hepatitis C with high dose consensus interferon induction therapy. Gastroenterology 124(4):A214.